CLINICAL TRIAL: NCT00882167
Title: Sensitivity and Predictive Value of Functional Cine Magnetic Resonance Imaging (MRI) Detecting Intra-abdominal Adhesions
Brief Title: Cine-magnetic Resonance Imaging (MRI) Detecting Intra Abdominal Adhesions
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: RU-RTB-0001
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Tissue Adhesions
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with laparotomy in history
  Interventions: Other: CineMRI

INTERVENTIONS:
Other: CineMRI — CineMRI scan of the abdomen at 1.5 Tesla.

SUMMARY:
Official title:

Sensitivity and predictive value of functional cine magnetic resonance imaging (MRI) detecting intra-abdominal adhesions

Background:

Adhesions are a frequent problem in abdominal surgery. The formation of adhesions is part of a normal wound healing. However in some patients adhesions cause severe complications such as chronic pain, obstruction and strangulation of the bowel. Adhesions can also obstruct access to the peritoneal cavity and complicate reoperations. Accurate imaging of adhesions would be of benefit avoiding adhesion related complications at repeated laparotomy or laparoscopy. At present no validated diagnostic tool mapping adhesions exists.

Purpose:

To define the sensitivity and specificity of functional cineMRI in detecting and mapping adhesions in patients undergoing reoperation.

Design:

Prospective multicenter observational trial

Primary outcome:

Sensitivity and specificity of functional MRI detecting adhesions to the abdominal wall

Secondary outcome:

Sensitivity and specificity of functional MRI detecting organ-to-organ adhesions.

Estimated enrollment: 100

Estimated study completion date: dec 2019

Estimated primary completion date: dec 2019

ELIGIBILITY:
Inclusion Criteria:

* Patients with a median abdominal scar due to a previous open abdominal surgical procedures with a length of at least 10 cm and have given written consent.

Exclusion Criteria:

* Severe claustrophobia.
* No MRI allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who will undergo elective abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-04; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity | 2 weeks
  diagnsotic accuracy for detecting adhesions

CONTACTS AND LOCATIONS:
Overall Officials: Harry van Goor, MD, PhD, Study Director — Radboud University Nijmegen Medical Center; Richard PG ten Broek, Principal Investigator — Radboud University Nijmegen Medical Center
Locations (5):
- Netherlands (5):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Radboud University Nijmegen Medical Center, Nijmegen, Gelderland
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Gelre Hospital, Apeldoorn
  - Catharina Hospital, Eindhoven

REFERENCES:
- [Background] van Goor H. Consequences and complications of peritoneal adhesions. Colorectal Dis. 2007 Oct;9 Suppl 2:25-34. doi: 10.1111/j.1463-1318.2007.01358.x. PMID 17824967
- [Background] Lienemann A, Sprenger D, Steitz HO, Korell M, Reiser M. Detection and mapping of intraabdominal adhesions by using functional cine MR imaging: preliminary results. Radiology. 2000 Nov;217(2):421-5. doi: 10.1148/radiology.217.2.r00oc23421. PMID 11058638
- [Background] Mussack T, Fischer T, Ladurner R, Gangkofer A, Bensler S, Hallfeldt KK, Reiser M, Lienemann A. Cine magnetic resonance imaging vs high-resolution ultrasonography for detection of adhesions after laparoscopic and open incisional hernia repair: a matched pair pilot analysis. Surg Endosc. 2005 Dec;19(12):1538-43. doi: 10.1007/s00464-005-0092-y. Epub 2005 Oct 24. PMID 16247569